CLINICAL TRIAL: NCT01112358
Title: Lutropin Alfa (Luveris®) in Women at Risk of Poor Response Suppressed With Cetrorelix: an Exploratory Trial
Brief Title: Lutropin Alfa in Women at Risk of Poor Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP26170 (INI25954); 2005-002229-30 (EudraCT Number)
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Stimulation
Keywords: Lutropin alfa; Fertilization in vitro; Intracytoplasmic sperm injection; Reproductive techniques, assisted
MeSH Terms: conditions — Helping Behavior | interventions — follitropin alfa; Luteinizing Hormone, beta Subunit; cetrorelix; Progesterone

ARMS (2):
- r-FSH + r-hLH (Experimental): Lutropin alfa (r-hLH) will be administered at a daily dose of 150 International Units (IU) from the presence of at least one follicle greater than (>) 14 millimeter (mm) to complete ovarian stimulation. Follitropin alfa (r-FSH) will be administered at an initial dose of 225-450 IU per day (according to standard center practice); the dose will then be adjusted to ovarian response as assessed by ovarian ultrasound and/or serum estradiol. Participants will also receive analogous GnRH antagonist and natural progesterone, as per standard center practice. To complete follicular maturation and trigger ovulation, a single dose of 250 milligrams (mg) of recombinant Human Chorionic Gonadotropin (r-hCG) will be administered subcutaneously at 12 hours after the last injection of lutropin alfa and/or follitropin alfa and analogous GnRH antagonist.
  Interventions: Drug: r-FSH; Drug: r-hLH; Drug: Analogous GnRH antagonist; Drug: r-hCG; Drug: Progesterone
- r-FSH (Active Comparator): Follitropin alfa (r-FSH) will be administered at an initial dose of 225-450 IU per day (according to standard center practice); the dose will then be adjusted to ovarian response as assessed by ovarian ultrasound and/or serum estradiol. Participants will also receive analogous GnRH antagonist and natural progesterone, as per standard center practice. To complete follicular maturation and trigger ovulation, a single dose of 250 mg of r-hCG will be administered subcutaneously at 12 hours after the last injection of follitropin alfa and analogous GnRH antagonist.
  Interventions: Drug: r-FSH; Drug: Analogous GnRH antagonist; Drug: r-hCG; Drug: Progesterone

INTERVENTIONS:
Drug: r-FSH — r-FSH will be administered as specified in the arm description.
  Other Names: Follitropin alfa; Gonal-F®
Drug: r-hLH — r-hLH will be administered as specified in the arm description.
  Other Names: Lutropin alfa; Luveris®
  Arms: r-FSH + r-hLH
Drug: Analogous GnRH antagonist — Analogous GnRH antagonist will be administered as specified in the arm description.
  Other Names: Cetrotide®
Drug: r-hCG — r-hCG will be administered as specified in the arm description.
Drug: Progesterone — Progesterone will be administered as specified in the arm description.

SUMMARY:
Evaluate the effectiveness of adding lutropin alfa (recombinant human luteinizing hormone [r-hLH]) in the middle of the follicular phase compared to no addition, in infertile women at risk of poor response stimulated with follitropin alfa (recombinant Follicle-Stimulating Hormone [r-FSH]) under Gonadotropin Releasing Hormone (GnRH) antagonist in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI), in the number and quality of oocytes, follicular development, fertilization oocyte, embryo quality, and pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were at risk of poor response by at least one of the following criteria: a) <3 follicles in last cycle, or less than or equal to (</=) 2 metaphase II oocytes, or estradiol (E2) <600 pg/mL; b) Cancellation of previous cycle; c) Early follicular serum Follicle-Stimulating Hormone (FSH) >8.5 milli IU/L
* Participants with normal baseline luteinizing hormone and E2 levels
* Regular menstrual cycles of 25-35 days
* Presence of both ovaries and uterus able to withstand pregnancy

Exclusion Criteria:

* Participants who had any clinically significant disease including known human immunodeficiency virus (HIV), hepatitis-B virus (HBV)/hepatitis-C virus (HCV) positivity
* Participants with more than 3 previous assisted reproductive techniques (ART) cycles
* Participants with polycystic ovaries or cyst of unknown etiology; unexplained gynecological bleeding
* Participants who had any contraindication to being pregnant
* Active substance abuse
* Participants who had simultaneously participated in another clinical drug trial

Max Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2005-12-07 (Actual); Primary Completion 2007-01-30 (Actual); Study Completion 2007-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Hospital Universitario de La Fe, Valencia, Spain

REFERENCES:
- [Result] M.J. Fernández Ramírez, A. Monzó, T. García-Gimeno, J.M. Rubio, V. Montañana, C. Duque, G. Herrero, A. Romeu. Role of LH administration during the follicullar phase in women with risk of low response in ovarian stimulation with FSH and cetrorelix for IVF, REVISTA IBEROAMERICANA DE FERTILIDAD, Vol. 23- nº 5 - Septiembre-Octubre 2006
- See also: Results publication in spanish language — http://www.revistafertilidad.org/RecursosWEB/fertilidad/Fertil%20Sept-oct-trab-1%2006.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- r-FSH + r-hLH: Lutropin alfa (recombinant human luteinizing hormone [r-hLH]) was administered at a daily dose of 150 International Units (IU) from the presence of at least one follicle greater than (>) 14 millimeter (mm) to complete ovarian stimulation. Follitropin alfa (recombinant Follicle-Stimulating Hormone [r-FSH]) was administered at an initial dose of 225-450 IU per day (according to standard center practice); the dose was then adjusted to ovarian response as assessed by ovarian ultrasound and/or serum estradiol. Participants also received analogous Gonadotropin Releasing Hormone (GnRH) antagonist and natural progesterone, as per standard center practice. To complete follicular maturation and trigger ovulation, a single dose of 250 milligrams (mg) of recombinant Human Chorionic Gonadotropin (r-hCG) was administered subcutaneously at 12 hours after the last injection of lutropin alfa and/or follitropin alfa and analogous GnRH antagonist (on Days 2 to 8).
- r-FSH: Follitropin alfa (r-FSH) was administered at an initial dose of 225-450 IU per day (according to standard center practice); the dose was then adjusted to ovarian response as assessed by ovarian ultrasound and/or serum estradiol. Participants also received analogous GnRH antagonist and natural progesterone, as per standard center practice. To complete follicular maturation and trigger ovulation, a single dose of 250 mg of r-hCG was administered subcutaneously at 12 hours after the last injection of follitropin alfa and analogous GnRH antagonist (on Days 2 to 8).
Period: Overall Study
Arm/Group | r-FSH + r-hLH | r-FSH
Started | 25 | 33
Completed | 25 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomly assigned to one of two treatment groups and received at least one dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | r-FSH + r-hLH | r-FSH | Total
Number analyzed (Participants) | 25 | 33 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (2.2) | 34.4 (2.0) | 34.65 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 33 | 58
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Time Frame: At the end of stimulation (Day 2 up to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Oocytes | 4.0 (5.3) | 3.5 (3.1)

2. Primary Outcome: Number of Follicles Greater Than (>) 14 Millimeter (mm) in Diameter
Time Frame: At the end of stimulation (Day 2 up to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Follicles | 7.2 (1.1) | 7.0 (0.8)

3. Primary Outcome: Oocytes Recovery Rate
Description: Oocytes recovery rate (oocytes per >14 mm follicle) is defined as number of oocytes retrieved divided by number of follicles >14 mm in diameter.
Time Frame: At the end of stimulation (Day 2 up to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: oocytes per >14 mm follicle
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
oocytes per >14 mm follicle | 0.56 (0.42) | 0.50 (0.41)

4. Secondary Outcome: Oocyte Nuclear Maturity Rate
Description: Oocyte nuclear maturity rate (metaphase II oocytes per retrieved oocyte) is defined as number of metaphase II oocytes divided by total number of oocytes retrieved.
Time Frame: At the end of stimulation (Day 2 up to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: metaphase II oocytes/retrieved oocyte
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
metaphase II oocytes/retrieved oocyte | 0.73 (0.75) | 0.61 (0.26)

5. Secondary Outcome: Fertilization Rate
Description: The fertilization rate (2 pronuclei [PN] fertilized oocytes per inseminated oocyte) was defined as number of 2 PN fertilized oocytes divided by number of inseminated oocytes.
Time Frame: Up to 35-45 days after administration of r-hCG (r-hCG administration = Day 2 to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: 2PN fertilized oocyte/inseminated oocyte
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
2PN fertilized oocyte/inseminated oocyte | 0.70 (0.35) | 0.64 (0.33)

6. Secondary Outcome: Number of Embryos by Quality
Description: Embryo quality was graded according to morphological classification of Veeck. Grade 1: even blastomeres with no fragmentation; Grade 2: even blastomeres with slight fragmentation (less than 20%); Grade 3: uneven size blastomeres with no fragmentation; Grade 4: even or uneven size blastomeres with moderate fragmentation (20-25%); and Grade 5: unrecognizable blastomeres with severe fragmentation (>50%).
Time Frame: Up to 35-45 days after administration of r-hCG (r-hCG administration = Day 2 to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Embroys
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Embroys
  Grade 1 | 0.6 (0.7) | 0.8 (1.0)
  Grade 2 | 1.4 (1.8) | 0.7 (0.76)
  Grade 3 | 1.8 (2.0) | 0.6 (0.8)
  Grade 4 | 0.1 (0.2) | 0.2 (0.3)
  Grade 5 | 0.1 (0.2) | 0.0 (0.2)

7. Secondary Outcome: Number of Embryos Transferred by In Vitro Fertilization (IVF)
Time Frame: Up to 35-45 days after administration of r-hCG (r-hCG administration = Day 2 to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Embroys
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Embroys | 2.0 (1.0) | 1.6 (0.8)

8. Secondary Outcome: Number of Participants With Positive Pregnancy Test
Description: The beta Human Chorionic Gonadotropin (beta-hCG) test was used as pregnancy test.
Time Frame: Up to 35-45 days after administration of r-hCG (r-hCG administration = Day 2 to Day 8)
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Participants | 3 | 5

9. Secondary Outcome: Number of Participants With Clinical Pregnancy
Description: A clinical pregnancy is a pregnancy that is confirmed by both pregnancy test (beta-hCG test) and sonographic confirmation of a gestational sac or heartbeat (fetal sac).
Time Frame: Up to 35-45 days after administration of r-hCG (r-hCG administration = Day 2 to Day 8)
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Participants | 3 | 5

10. Secondary Outcome: Implementation Rate
Description: Implementation rate (clinical pregnancy/embryo transferred) was defined as the number of clinical pregnancies divided by number of embryos transferred.
Time Frame: Up to 35-45 days after administration of r-hCG (r-hCG administration = Day 2 to Day 8)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Clinical pregnancy/embryo transferred
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Clinical pregnancy/embryo transferred | 0.15 [0.05 to 0.33] | 0.14 [0.05 to 0.28]

11. Secondary Outcome: Plasma Level of Estradiol
Time Frame: At the time of r-hCG administration (any days between Day 2 to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Picograms per milliliters (pg/mL)
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Picograms per milliliters (pg/mL) | 1218 (699) | 1029 (336)

12. Secondary Outcome: Endometrial Thickness
Time Frame: At the time of r-hCG administration (any days between Day 2 to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
millimeters (mm) | 12.3 (1.8) | 11.2 (2.1)

13. Secondary Outcome: Duration of Ovarian Stimulation
Description: Duration of ovarian stimulation was defined as the time from start of study treatment to time of r-hCG administration.
Time Frame: Randomization to Day 8
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
days | 4.8 (1.7) | 4.8 (1.7)

14. Secondary Outcome: rFSH Cumulative Dose
Time Frame: Randomization to Day 8
Population: ITT population
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
IU | 4338 (1241) | 4298 (1137)

15. Secondary Outcome: Plasma Levels of LH
Time Frame: At the time of r-hCG administration (any days between Day 2 to Day 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: IU per liter (IU/L)
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
IU per liter (IU/L) | 2.8 (1.0) | 2.1 (2.1)

16. Secondary Outcome: Number of Participants in Whom At Least 1 Stimulation Cycle Was Cancelled
Time Frame: Randomization to Day 8
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | r-FSH + r-hLH | r-FSH
Number analyzed (Participants) | 25 | 33
Participants | 8 | 8

ADVERSE EVENTS:
Arm/Group | r-FSH + r-hLH | r-FSH
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/33
Other Adverse Events (participants affected / at risk) | 0/25 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No